CLINICAL TRIAL: NCT05742113
Title: DYSPNEA: PERFUSION INDEX and TRIAGE STATUS (the Name of the Project)
Brief Title: Emergency Classification According to Fingertip Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manisa Celal Bayar University (Other)
Responsible Party: Principal Investigator, Cumhur Murat TULAY, Aaa.Prof., Manisa Celal Bayar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10.10.2018 and 20.478.486; Manisa Celal Bayar University (Other: 2018-213)
Record Dates: First submitted 2023-01-31; First posted 2023-02-23 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dyspnea
Keywords: Dyspnea; Emergency; Perfusion index; Triage
MeSH Terms: conditions — Dyspnea; Emergencies

STUDY DESIGN:
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Triage status red (Experimental): the relationship between the perfusion index and the emergency triage classification in patients admitted to the emergency department with dyspnea.
  Interventions: Device: Masimo Radical-7

INTERVENTIONS:
Device: Masimo Radical-7 — perfusion index measuring device

SUMMARY:
Dyspnea is one of the most common reasons for admission to the emergency department[1]. Oxygen saturation has great importance in determining the triage status of patients admitted to the hospital with dyspnea and planning the emergency treatment [2].

Peripheral perfusion index (PI), which shows tissue oxygenation is a noninvasive way of demonstrating tissue perfusion in critically ill patients. Studies have shown that PI is an accurate, fast and reliable pulse oximetry-based indicator of tissue perfusion [3-5]. PI shows the perfusion status of the tissue in the applied area for an instant and a certain time interval. The PI value ranges from 0.02% (very weak) to 20% (strong) [6].

Triage scales are used to distinguish emergency and non-emergency patients. The emergency triage system is used to quickly determine the care priorities of patients during admission to the emergency department[7,8].

It is important to make the triage classification for dyspnea in emergency services quickly and accurately to start the treatment protocols as early as. In this study, the investigators aimed to determine the relationship between perfusion index and the emergency triage classification in patients admitted to the emergency department with dyspnea.

DETAILED DESCRIPTION:
Purpose: To determine the effect of PI measurement on the emergency triage classification in patients with dyspnea.

Methods: Adult patients who presented with dyspnea and whose perfusion index values were measured with Masimo Radical-7 device at the time of admission, at the first hour and the second hour of admission were included in the study. The PI and oxygen saturation measured by finger probes were compared and the superiority of their effects on the emergency triage classification was compared.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over the age of 18 who presented with dyspnea
* whose perfusion index values were measured at the time of first admission (arrival time), at the first hour and the second hour of admission were included in the study

Exclusion Criteria:

* Patients who applied due to the mechanism of trauma,
* patients with known vascular disease (Buerger's disease, peripheral artery disease, etc.), -patients with COVID-19 PCR positivity
* whose perfusion index measurement could not be completed due to hospitalization or discharge were excluded from the study.

Ages: 18 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1490 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Perfusion index use for triage status | perfusion index measurement at the time of first admission to hospital
  for determination of triage status of patients with dyspnea with using perfusion index
Perfusion index use for triage status | perfusion index measurement at the time of the first hour after admission to hospital
  for determination of triage status of patients with dyspnea with using perfusion index
Perfusion index use for triage status | perfusion index measurement at the time of the second hour after admission to hospital
  for determination of triage status of patients with dyspnea with using perfusion index

CONTACTS AND LOCATIONS:
Overall Officials: Cumhur M TULAY, Ass.Prof., Principal Investigator — Ass.Prof.
Locations (1):
- Manisa Celal Bayar University, Manisa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The result will be explained in the manuscript when published.